CLINICAL TRIAL: NCT03223649
Title: Break It Up: A Study Evaluating Breaking Up Daily Sedentary Behavior in Youth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 170130; 17-CH-0130 (Other: NIH Clinical Center - protocol number)
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-01-04

CONDITIONS: Healthy; Obesity; Overweight
Keywords: Metabolism; Children; Walking Bouts; Glucose; Insulin
MeSH Terms: conditions — Obesity; Overweight; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentary (Experimental): (Control intervention) Six daily 3 hour sessions with no physical activity (i.e. subject remains sedentary in seated or recumbent position) throughout the 3 hour duration.
  Interventions: Other: Sedentary
- Walking bouts (Experimental): Six daily 3 hour sessions with prompted 3-minute moderate-intensity walking bouts performed on a treadmill every 30 minutes throughout the 3 hour duration. There will be a total of 6 walking bouts (18 minutes total) each day. Moderate-intensity walking speed and grade will be selected to achieve 80% of the heart rate achieved at the ventilatory threshold as determined during a V02max test.
  Interventions: Other: Walking Bouts

INTERVENTIONS:
Other: Walking Bouts — Six daily 3 hour sessions with prompted 3-minute moderate-intensity walking bouts performed on a treadmill every 30 minutes throughout the 3 hour duration. There will be a total of 6 walking bouts (18 minutes total) each day. Moderate-intensity walking speed and grade will be selected to achieve 80% of the heart rate achieved at the ventilatory threshold as determined during a V02max test.
  Arms: Walking bouts
Other: Sedentary — (Control 'intervention') Six daily 3 hour sessions with no physical activity (i.e. subject remains sedentary in seated or recumbent position) throughout the 3 hour duration.
  Arms: Sedentary

SUMMARY:
Background:

Some studies have found that people can better process sugars when they take walking breaks. Studies have also found that children's attention and memory may improve after exercise. It is not known if short walking breaks have the same effects. Researchers want to study if breaking up sitting with walking for 6 days helps children s bodies use sugars and improves concentration.

Objectives:

To learn if breaking up sedentary (low-activity) time with short walking breaks over 6 days affects how children s bodies use sugar. To learn if breaking up sedentary time changes children s attention, memory, feelings, activity, or eating.

Eligibility:

Children ages 7-11 in general good health

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Fasting blood tests. On 2 out of 7 total study visits, participants cannot eat or drink after 10 p.m. the night before.
* Full-body X-ray
* EKG (Electronic signals that record heart function through stickers)
* Treadmill exercise. Heart, blood pressure, and oxygen will be monitored.
* Questions about the child s health, socialization, and activity, and parent s education and economic status
* Picture vocabulary test
* Dietician meeting (Questions about eating habits)

Participants will have visits on 6 consecutive days. Over that time, they will wear 2 devices to monitor blood sugar and activity (even while at home).

Participants will have 5 after-school visits. These include:

* Health check
* Snack plus food for the next 24 hours
* Activity monitored
* 3-hour sitting tests. Participants will do non-active things. Some will have 3-minute walks every 30 minutes.
* Cognitive tests and questions about mood and anxiety are given on days #1 & 5.

Participants will fast before the last visit in the morning. They will have:

* 9 blood draws by IV catheter. Participants will drink sugar water.
* Sitting test
* Activity monitored
* Meal (food buffet)

DETAILED DESCRIPTION:
Background:

Sedentary behavior is defined as a set of low-intensity activities involving limited body movement (e.g.: TV viewing, prolonged sitting). Some studies have found higher levels of childhood sedentary behavior predict higher body mass index (BMI) and metabolic abnormalities. We and others have found that interrupting sitting with short, 2-3 minute bouts of moderate activity (walking) can improve glucose tolerance during a single session. Thus, interrupting sedentary behavior may be an intervention strategy to reduce health risks.

Objective:

We propose to conduct a randomized pilot study to assess whether interrupting sedentary behavior for 6 consecutive days provides sustained improvement in carbohydrate metabolism without negatively impacting executive function, attention, mood, anxiety, dietary

intake or usual physical activity.

Design & Population:

Using a randomized parallel group design, children, ages 7-11 years, will complete an assigned randomized condition of either 6 consecutive days of 3 hours of monitored sedentary activity (sitting) or 6 consecutive days of 3 hours of interrupted sitting (in which they will be prompted to walk for 3 minutes every 30 minutes).

Outcome measures:

Twenty-four-hour continuous glucose monitoring and postprandial insulin incremental area under the curve (iAUC) on post-condition oral glucose tolerance testing will be the primary measures. Secondary measures include: postprandial glucose iAUC, executive function, attention, mood, anxiety, dietary intake, and free-living physical activity.

Impact:

This project will investigate if consecutive daily interruption of sitting behaviors improves glucose tolerance, a potential negative health consequences of sedentary behavior in children. If repeatedly interrupting sitting with short bouts has sustained beneficial effects among children, interventions examining the frequency, duration, and intensity of such interruptions could be developed for use in the community setting. Thus, these results have the potential to provide insight into novel behavioral intervention targets in youth.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will qualify for the study if they meet the following criteria:

1. Good general health.
2. Age greater than or equal to 7 and less than 12 years.
3. Fasting plasma glucose less than 100 mg/dL
4. Body mass index (BMI) greater than or equal to the 5th percentile, as determined by the CDC age- and sex- specific growth charts.

EXCLUSION CRITERIA:

Participants will be excluded from the study for:

1. Significant cardiac or pulmonary disease likely to or resulting in hypoxia or decreased perfusion.
2. Evidence of impaired glucose tolerance or type 2 diabetes, including fasting plasma glucose greater than or equal to 100 mg/dL.
3. Presence of other endocrinologic disorders leading to obesity (e.g.: Cushing Syndrome).
4. Participants who have, or whose parent/guardians have, current substance abuse or a psychiatric disorder or other condition that, in the opinion of the investigators, would impede competence, compliance, or prevent the completion of the study.
5. Participants who have, or are currently receiving, anti-psychotic drugs that would affect metabolism, cognitive outcomes, and body habitus.
6. Participants receiving medical treatment other than diet for hypertension or dyslipidemia.
7. Participants with precocious puberty and/or receiving androgen and estrogen therapy.
8. Participants currently taking medications for ADHD, or any disorder or use of medications known to affect body composition or weight including but not limited to glucocorticoids or other steroid compounds.
9. Presence of pre-existing neurocognitive disabilities, or an age-adjusted score below 85 on the Picture Vocabulary Test at the screening visit.
10. Presence of food allergies, such as peanut/tree nut, dairy, soy or any other food allergy or personal dietary restrictions that would preclude participant from consuming the daily diet or the buffet.
11. Presence of significant skin disease or allergy to adhesive material prohibiting placement of a continuous glucose monitor.
12. Participants unable or unwilling to abstain from acetaminophen, ascorbic acid, or salicylic acid during study duration.
13. Participant does not speak fluent English.
14. Participant is or becomes pregnant.
15. Participant has an ambulatory impairment

OPTIONAL MRS SUPPLEMENTAL ARM

INCLUSION CRITERIA

(a) Participants will qualify for the study if they qualify for the primary Break It Up! study.

EXCLUSION CRITERIA

1. Cannot have MRI scanning. Some of the reasons a child might not be able to have MRI include:

   * Implanted cardiac pacemaker or defibrillator
   * Cochlear Implants
   * Ocular foreign body (e.g. metal shavings)
   * Embedded shrapnel fragments
   * Central nervous system aneurysm clips
   * Implanted neural stimulator
   * Medical infusion pumps
   * Any implanted device that is incompatible with MRI.
2. Is not likely to tolerate an MRI scan. Examples of medical conditions that would make it difficult to undergo MRI include severe anxiety (nervousness) or hyperactivity which make it hard for your child to lay flat for the study.
3. Requires sedation for MRI studies.
4. Has a condition that makes entry into the scanner difficult (e.g. weight over 550 lbs, claustrophobia, etc.).
5. Has severe back-pain or motion disorders that make it hard for a child to lie on his/her back within the MRI scanner and hold still for the scan.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2021-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual level deidentified data for all sociodemographic characteristics and outcomes will be made available after publication of the study primary outcome.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication of the primary outcome for 5 years
Access Criteria: A data sharing agreement may have to be negotiated with NICHD. Contact Dr. Jack Yanovski jy15i@nih.gov, 301-496-0858.

REFERENCES:
- [Background] Broadney MM, Belcher BR, Berrigan DA, Brychta RJ, Tigner IL Jr, Shareef F, Papachristopoulou A, Hattenbach JD, Davis EK, Brady SM, Bernstein SB, Courville AB, Drinkard BE, Smith KP, Rosing DR, Wolters PL, Chen KY, Yanovski JA. Effects of Interrupting Sedentary Behavior With Short Bouts of Moderate Physical Activity on Glucose Tolerance in Children With Overweight and Obesity: A Randomized Crossover Trial. Diabetes Care. 2018 Oct;41(10):2220-2228. doi: 10.2337/dc18-0774. Epub 2018 Aug 6. PMID 30082324
- [Background] Belcher BR, Berrigan D, Papachristopoulou A, Brady SM, Bernstein SB, Brychta RJ, Hattenbach JD, Tigner IL Jr, Courville AB, Drinkard BE, Smith KP, Rosing DR, Wolters PL, Chen KY, Yanovski JA. Effects of Interrupting Children's Sedentary Behaviors With Activity on Metabolic Function: A Randomized Trial. J Clin Endocrinol Metab. 2015 Oct;100(10):3735-43. doi: 10.1210/jc.2015-2803. Epub 2015 Aug 27. PMID 26312582
- [Background] Dunstan DW, Kingwell BA, Larsen R, Healy GN, Cerin E, Hamilton MT, Shaw JE, Bertovic DA, Zimmet PZ, Salmon J, Owen N. Breaking up prolonged sitting reduces postprandial glucose and insulin responses. Diabetes Care. 2012 May;35(5):976-83. doi: 10.2337/dc11-1931. Epub 2012 Feb 28. PMID 22374636
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-CH-0130.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via multiple methods:
  1. Letters were mailed to local parents
  2. Flyers were posted with permission.
  3. Local community groups were asked to send the flyer to their listservs.
  4. Schools, churches, pediatricians, and community centers were contacted.
  5. Potential volunteers in ResearchMatch program were contacted.
Pre-assignment Details: Of the 129 participants who were evaluated with baseline screening, 20 were not studied further:
  * 12: Failed to meet inclusion criteria
    * 2: Impaired glucose tolerance
    * 1: Hepatic disease
    * 7: Failed picture vocabulary test
    * 2 Did not meet BMI criteria
  * 6: No longer interested
  * 1: Could not determine VO2 max or lactate threshold from exercise testing (insufficient effort)
  * 1: Withdrawn due to COVID pandemic restrictions
Groups:
- Walking Bouts: Six daily 3 hour sessions with prompted 3-minute moderate-intensity walking bouts performed on a treadmill every 30 minutes throughout the 3 hour duration. There will be a total of 6 walking bouts (18 minutes total) each day. Moderate-intensity walking speed and grade will be selected to achieve 80% of the heart rate achieved at the ventilatory thresholdas determined during a V02max test.
  Walking Bouts: Six daily 3 hour sessions with prompted 3-minute moderate-intensity walking bouts performed on a treadmill every 30 minutes throughout the 3 hour duration. There will be a total of 6 walking bouts (18 minutes total) each day. Moderate-intensity walking speed and grade will be selected to achieve 80% of the heart rate achieved at the ventilatory threshold as determined during a V02max test.
Period: Overall Study
Arm/Group | Sedentary | Walking Bouts
Started | 52 | 57
Completed | 42 | 51
Not Completed | 10 | 6

BASELINE CHARACTERISTICS:
Population: Participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Sedentary | Walking Bouts | Total
Number analyzed (Participants) | 42 | 51 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (1.3) | 10.0 (1.2) | 10.2 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 24 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 36 | 43 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 27 | 38 | 65
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 51 | 93
Fat Mass (kg) [Mean (Standard Deviation); unit: kg] | 16.2 (12.4) | 13.5 (6.9) | 14.7 (9.8)
Lean Mass (kg) [Mean (Standard Deviation); unit: kg] | 28.9 (7.9) | 25.5 (4.8) | 27.0 (6.6)
Height (cm) [Mean (Standard Deviation); unit: cm] | 146.0 (9.8) | 141.2 (8.5) | 143.4 (9.4)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] — Weight in kg divided by the height, in meters, squared
  kg/m2 | 21.2 (6.6) | 19.9 (3.9) | 20.5 (5.3)
BMI z-score [Mean (Standard Deviation); unit: z-score] — The BMI Z-score indicates the number of standard deviations away from the mean BMI for age and sex. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population US National Standards for boys and girls from the Centers for Disease Control, which employs the LMS method for determining the Z-score
  z-score | 0.8 (1.2) | 0.8 (0.9) | 0.8 (1.0)
Fasting glucose (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 87.6 (6.8) | 87.9 (5.9) | 87.8 (6.3)
Fasting insulin (mIU/ml) [Mean (Standard Deviation); unit: mIU/mL] | 11.1 (9.8) | 9.7 (5.9) | 10.4 (7.4)
Peak VO2 (ml/kg/min) [Mean (Standard Deviation); unit: ml/kg/min] — Peak oxygen consumption per kg body weight per minute during an exercise test.
  ml/kg/min | 38.3 (9.1) | 38.5 (7.4) | 38.4 (8.1)
IPAQ score [Mean (Standard Deviation); unit: units on a scale (1-4)] — Average physical activity level within the previous 7 days reported on a questionnaire
  1. = Sedentary (less than 30 minutes of sustained activity a day, or <3.5 hours a week)
  2. = Low Active (30-45 minutes of sustained activity a day, or 3.5-5.25 hours a week)
  3. = Active (>45-90minutes of sustained activity a day, or >5.25-10.5 hours a week)
  4. = Very Active (>90 minutes of sustained activity a day, or >10.5 hours a week)
  units on a scale (1-4) | 2.2 (1.0) | 2.2 (1.1) | 2.2 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Insulin iAUC Obtained During the Oral Glucose Tolerance Test at the Final Experimental Visit.
Description: Insulin integrated area under the curve (iAUC) as a marker of glucose metabolism on OGTT during test day #6, collected at 0, 30, 60, 90, 120, 150, and 180 minutes after oral dextrose ingestion
Time Frame: test day 6
Measure: Mean (Standard Deviation); unit: mIU/dL∙min
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 42 | 51
mIU/dL∙min | 13,698.60 (9414.9) | 10,619.70 (6,781.30)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p = 0.005, ANCOVA — Unadjusted p-value; Log-transformed value adjusted for: arcsine sqrt transformed % fat mass, pubertal stage (pre, early, or late), and basal analyte log transformed; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-.17 to -.03], Standard Error of Mean .035

2. Secondary Outcome: Glucose iAUC Obtained During the Oral Glucose Tolerance Test on Day # 6 of Intervention.
Description: Integrated area under the curve (iAUC) for glucose values during the oral glucose tolerance test, collected at 0, 30, 60, 90, 120, 150, and 180 minutes after oral dextrose ingestion
Time Frame: test day 6
Measure: Mean (Standard Deviation); unit: mg/dL∙min
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 42 | 51
mg/dL∙min | 22,247.90 (2,927.70) | 21,688.80 (2,473.70)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p = 0.349, ANCOVA — Unadjusted P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.011, 95% CI 2-sided [-.033 to 0.011], Standard Error of Mean .011

3. Secondary Outcome: C-Peptide iAUC Obtained During the Oral Glucose Tolerance Test on Day # 6 of Intervention.
Description: Integrated area under the curve (iAUC) for C-Peptide values during the oral glucose tolerance test, collected at 0, 30, 60, 90, 120, 150, and 180 minutes after oral dextrose ingestion
Time Frame: test day 6
Measure: Mean (Standard Deviation); unit: ng/dL∙min
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 42 | 51
ng/dL∙min | 1,292.10 (449.8) | 1,160.10 (448.8)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p = .045, ANCOVA — Unadjusted p-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.043, 95% CI 2-sided [-.084 to -.002], Standard Error of Mean .021

4. Secondary Outcome: Free Fatty Acid iAUC Obtained During the Oral Glucose Tolerance Test on Day # 6 of Intervention.
Description: Integrated area under the curve (iAUC) for Free Fatty Acid values during the oral glucose tolerance test, collected at 0, 30, 60, 90, 120, 150, and 180 minutes after oral dextrose ingestion
Time Frame: test day 6
Measure: Mean (Standard Deviation); unit: mmol/L∙min
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 42 | 51
mmol/L∙min | 39.7 (9.8) | 38.5 (13.1)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p = 0.226, ANCOVA — Unadjusted p-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.019, 95% CI 2-sided [-0.051 to 0.013], Standard Error of Mean 0.016

5. Secondary Outcome: Daily Physical Activity (Step Counts/Min) During Intervention.
Description: Mean 3-dimensional activity during the 3 hours of intervention from all days (step counts per minute)
Time Frame: test days 1-6
Population: Data were unavailable from two participants randomized to the Sedentary condition and from one participant randomized to the Walking Bouts condition.
Measure: Mean (Standard Deviation); unit: step count per minute
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 40 | 50
step count per minute | 5.4 (1.9) | 11.2 (3.0)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -5.8, 95% CI 2-sided [-6.884 to -4.716], Standard Error of Mean 0.545

6. Secondary Outcome: Daily Physical Activity (3-dimensional Activity Counts/Day) Outside of the Intervention.
Description: Mean total daily 3-dimensional activity counts during the 21 hours without intervention on days 1-6 (activity counts/21 hours) from triaxial write accelerometers worn at home. Note: these are not "step counts" but total 3D activity counts because motion of the wrist at times other than walking are also recorded. There is no simple way to convert these counts to step counts.
Time Frame: test days 1-6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: activity counts per 21 hours x 10^6
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 40 | 50
activity counts per 21 hours x 10^6 | 2.1 (0.6) | 2.2 (0.5)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p = 0.39, t-test, 2 sided; Mean Difference (Final Values) = -0.100, 95% CI 2-sided [-0.330 to 0.130], Standard Error of Mean 0.116

7. Secondary Outcome: Energy Intake at the Final Test Meal.
Description: Total energy intake (kcal) during buffet meal immediately after the end of intervention
Time Frame: test day 6
Population: Data were unavailable from two participants randomized to the Sedentary condition and from two participants randomized to the Walking Bouts condition.
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 40 | 49
kcal | 1,312.4 (478.4) | 1,207.4 (443.8)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p = 0.648, ANCOVA; Dependent variable in Kcal log transformed, comparison adjusted for: age(y), lean mass(kg), fat mass(kg); Mean Difference (Final Values) = .021, 95% CI 2-sided [-0.071 to 0.114], Standard Error of Mean .046

8. Secondary Outcome: Percentage Fat Intake at the Final Test Meal.
Description: Percentage Energy intake from Fat during buffet meal immediately after the end of intervention
Time Frame: test day 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of total energy intake (%)
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 40 | 49
percentage of total energy intake (%) | 35.8 (7.0) | 36.2 (6.0)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p = 0.539, ANCOVA; Adjusted for age (years); Mean Difference (Final Values) = 0.834, 95% CI 2-sided [-1.857 to 3.525], Standard Error of Mean 1.354

9. Secondary Outcome: Percentage Carbohydrate Intake at the Final Test Meal.
Description: Percentage Energy intake from Carbohydrate during buffet meal immediately after the end of intervention
Time Frame: test day 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of total energy intake (%)
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 40 | 49
percentage of total energy intake (%) | 52.0 (9.0) | 51.8 (8.4)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p = 0.550, ANCOVA; Adjusted for age (years); Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-4.57 to 2.45], Standard Error of Mean 1.766

10. Secondary Outcome: Percentage Protein Intake at the Final Test Meal.
Description: Percentage Energy intake from Protein during buffet meal immediately after the end of intervention
Time Frame: test day 6
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percentage of total energy intake (%)
Arm/Group | Sedentary | Walking Bouts
Number analyzed (Participants) | 40 | 49
percentage of total energy intake (%) | 12.2 (3.6) | 12.0 (3.2)
Statistical Analysis 1: Comparison: Sedentary vs Walking Bouts; Test type: Superiority; p = 0.741, ANCOVA; Adjusted for age (years); Mean Difference (Final Values) = 0.226, 95% CI 2-sided [-1.127 to 1.579], Standard Error of Mean 0.681

ADVERSE EVENTS:
Time Frame: Days 1-6
Description: Standard clinicaltrials.gov definitions were used.
Arm/Group | Sedentary | Walking Bouts
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/51
Other Adverse Events (participants affected / at risk) | 0/42 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT03223649/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT03223649/ICF_001.pdf